CLINICAL TRIAL: NCT06013982
Title: Impact of a Structured Anxiety Reduction Program on Anxiety in Patients Who Are Discharged to Home Following an Acute Stroke in an Academic Medical Center
Brief Title: Stroke and Anxiety Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-00759
Record Dates: First submitted 2023-08-23; First posted 2023-08-28 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients discharged following acute care stroke (Experimental): Participation will last 3 months from enrollment. Demographic data will be retrieved from the electronic health record and the Generalized Anxiety Disorder-7 (GAD-7) Anxiety Questionnaire will be administered at baseline. Participants will repeat the GAD-7 in 3 months and an additional qualitative survey on their experience including an evaluation of the structured anxiety reduction program.
  Interventions: Behavioral: Anxiety Reduction Bundle

INTERVENTIONS:
Behavioral: Anxiety Reduction Bundle — The Anxiety Reduction Bundle intervention comprises the following resources:
  * Stroke Support Group
  * Anxiety Reduction Sheet
  * Understanding Anxiety Disorder sheet
  * Your body's response to anxiety sheet
  * Relaxation Tip sheet
  * Breathing Tip sheet and video
  * A sigh of Relief video

SUMMARY:
The purpose of this pilot study is to explore the impact that a structured anxiety reduction intervention program has on patients being discharged to home following an acute stroke in an academic medical center. Eligible participants will be screened and recruited by the research team through daily rounds. After completing the informed consent process, the research team will pull demographic information from the electronic health record (EHR) and REDCAP that includes ethnicity and support system. Participants will complete the Anxiety Screen Questionnaire (GAD-7 ANXIETY SURVEY) and will be provided with information regarding stroke support groups available with additional NYU Langone Health and the American Heart Association internet-based information regarding anxiety reduction (NYU Langone Health Anxiety Reduction Bundle). The participants will be encouraged to attend a stroke support group for 3 months and utilize the NYU Langone Health Anxiety Reduction Bundle provided. At the completion of the intervention (3 months), participants will be provided with the GAD-7 ANXIETY SURVEY again and a survey that includes open-ended questions and a program evaluation by email. Analysis will occur after final data is collected.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with an acute stroke
* Able to speak, read and write in English
* Not cognitively impaired, as per standard of care documentation in the EHR regarding mental status.
* Discharged to home
* Internet access including email
* Willingness to participate in an anxiety reduction program
* Length of hospital stay less than 5 days from the initial presentation of stroke symptoms
* Must be medically stable

Exclusion Criteria:

* Not diagnosed with an acute stroke
* Unable to speak, read and write in English as this intervention is not available in other languages and at this time, funding is not available in order to have the resources provided translated or to have translation services available for these participants.
* Not discharged to home
* No internet access including email
* Unwilling or unable to participate in an anxiety reduction program
* Cognitively impaired
* Length of hospital stay greater than 6 days from the initial presentation of stroke symptoms
* Not medically stable

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Change in GAD-7 Score from Baseline to Month 3 | Baseline, Month 3
  The GAD-7 Anxiety Questionnaire involves 7 items assessing how often participants have felt bothered by anxiety-related problems over the past two weeks. Each item is rated on a Likert scale from 0 (not at all) to 3 (nearly every day). The total score is the sum of responses and ranges from 0-21; where 0-4 = minimal anxiety; 5-9 = mild anxiety; 10-14 = moderate anxiety; 15-21 = severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Bibi Sangster, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot study and the data will need to be evaluated before it is shared.